CLINICAL TRIAL: NCT07272837
Title: GLP-1 Receptor Agonist-Induced Loss and Impairment of Muscle Mass - Evaluation of Response
Brief Title: Impact of Semaglutide (Ozempic/Wegovy®) on Heart and Muscle Mass
Acronym: GLIMMER
Status: Not yet recruiting | Type: Observational
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00153724
Record Dates: First submitted 2025-11-26; First posted 2025-12-09 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Type 2 Diabetes; Obesity; Semaglutide
Keywords: Semaglutide; Type 2 Diabetes; Diabetes; Obesity; Body Composition; Muscle Mass; Skeletal Muscle Mass; Cardiac Muscle Mass; GLP-1 Receptor Agonist
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — If a participant consents, their blood samples will be retained for up to 10 years after the completion of the main study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to use advanced MRI scans to track changes in both muscle and fat in the body and heart over a 12-month period in individuals starting semaglutide. By doing so, we hope to gain a clearer understanding of how semaglutide affects muscle health and function. Our goal is to ensure the medication supports long-term well-being, particularly for people who may be at higher risk of muscle loss.

This study involves (3) in-person study visits. At each visit, participants will be asked to:

* Undergo magnetic resonance imaging (MRI) while resting and during exercise to take pictures of their heart, abdomen, and legs.
* Complete tests to assess balance, sit-to-stand, walking speed, and handgrip strength.
* Complete questionnaires (related to demographics, health information, physical activity, and nutrition).
* Have a blood sample collected.
* Have blood ketone levels assessed through two finger pricks.
* Complete three days of food records.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18-75 years of age
* Starting semaglutide for type 2 diabetes or weight loss (body mass index ≥27.5kg/m2)
* Able to safely undergo an MRI scan (including meeting the physical requirements for MRI equipment)

Exclusion Criteria:

* Current use of semaglutide for more than 2 weeks
* Major recent heart issues or other severe health conditions
* Concerns related to MRI use (including metal implants, pacemaker, severe claustrophobia)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Residents of Edmonton, AB or the surrounding area who are able to attend study visits at the Mazankowski Alberta Heart Institute.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Changes in skeletal and cardiac muscle mass | 12 months

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study information and pre-screening survey — https://redcap.link/glimmer